CLINICAL TRIAL: NCT02186236
Title: A Pilot Study Testing the Detection of Oncogenic Tumor Mutations in the Urine and Blood of Lung and Colorectal Cancer Patients
Brief Title: Detection of Oncogenic Tumor Mutations in the Urine and Blood of Lung and Colorectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Cardiff Oncology (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-114
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Lung Cancer; Colorectal Cancer
Keywords: Detection of Oncogenic Tumor Mutations; blood; urine; 14-114
MeSH Terms: conditions — Lung Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — periphera blood sample and urine sample

GROUPS / COHORTS (1):
- Lung and Colorectal cancer patients: Eligible people who consent to participation will provide urine (both in lung cancer and colorectal cancer) and blood (in lung cancer only) samples at pre-specified times.

SUMMARY:
The purpose of this study is to see whether gene mutations can be found in the urine or blood of lung cancer patients and urine of colorectal cancer patients. Gene mutations are when DNA in a gene is damaged in a way that changes the genetic message carried by that gene. Gene mutations can sometimes cause lung cancers. These gene mutations are only found in lung and colorectal cancer cells, not the normal cells in your body. All lung cancer tumors and colorectal cancer tumors are now tested for different gene mutations as their presence affects lung cancer treatment. Tumor samples obtained from a biopsy or surgery are typically tested for these gene mutations.

ELIGIBILITY:
Inclusion Criteria:

Lung cancer:

For patients participating in Part A (initial testing) and Part B (serial testing):

* Patients must have a diagnosis of stage IV lung adenocarcinoma undergoing systemic therapy.
* Patients must have had or intend to have EGFR mutation testing (specifically including exon 19 deletions and L858R) performed on their tumor with results available from a CLIA certified laboratory.
* ≥ 18 years of age

Specific to patients participating in Part B (serial testing):

* Patients must be planning to receive cancer care at Memorial-Sloan Kettering.
* Patients must have a confirmed EGFR mutant lung cancer (exon 19 deletions and L858R) with molecular testing results available from a CLIA certified laboratory.
* Must be within 3 months of their diagnosis of metastatic lung cancer.
* Treatment plan should include an EGFR tyrosine kinase inhibitor, but may concurrently be on a therapeutic protocol.

Colorectal Cancer:

For patients participating in Part A (initial testing) and Part B (serial testing):

* Patients must have a diagnosis of stage IV colorectal adenocarcinoma undergoing systemic therapy or have recently progressed on therapy including anti-EGFR based therapy.
* Patients must have had or intend to have RAS/RAF mutation testing on their tumor with results available from a CLIA certified laboratory. For the patients who recently progressed on anti-EGFR must have tumor tissue molecular analyses preformed (prior to enrolling or a plan to test it at the time of enrollment).
* >18 years of age

Specific to patients participating in Part B (serial testing):

* Patients must be planning to receive cancer care at Memorial-Sloan Kettering.
* Patients must have a confirmed RAS/RAF mutant colorectal cancer with molecular testing results available from a CLIA certified laboratory.
* Must be within 3 months of their diagnosis of metastatic colorectal cancer.

Exclusion Criteria:

lung cancer and colorectal cancer

* Comorbidities that would prohibit or make serial urine collection difficult or impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC clinics
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2014-07; Primary Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
EGFR detection in urinary cell free DNA [cfDNA] | 2 years
  The Trovagene urine-based assay will test to determine the presence of EGFR mutation in cfDNA or RAS/RAF mutation in colorectal cancer
To validate the Trovagene urine assay | 2 years
  urine assay to identify EGFR mutations as compared to the gold standard of tumor tissue.

SECONDARY OUTCOMES:
EGFR detection in plasma circulating tumor cells [CTC] and plasma cfDNA) | 2 years
  The plasma-based assay will test to determine the presence of EGFR mutation in CTC and in cfDNA.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Yu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering West Harrison, East White Plains, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center at Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/